CLINICAL TRIAL: NCT02607618
Title: A Phase 3, Randomized, Double-blind, Multicenter Study to Evaluate the Safety and Efficacy of Intravenous Iclaprim Versus Vancomycin in the Treatment of ABSSSI: REVIVE-2
Brief Title: Phase 3 Study to Evaluate Safety and Efficacy of Iclaprim Versus Vancomycin for ABSSSI: REVIVE-2
Acronym: REVIVE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Motif Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICL-24-ABSSSI2
Record Dates: First submitted 2015-11-13; First posted 2015-11-18 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-06

CONDITIONS: Skin Structures and Soft Tissue Infections
MeSH Terms: conditions — Soft Tissue Infections | interventions — iclaprim; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- iclaprim (Experimental): iclaprim 80 mg intravenous every 12 hours
  Interventions: Drug: Iclaprim
- vancomycin (Active Comparator): vancomycin 15 mg/kg intravenous every 12, 24 or 48 hours based on creatinine clearance
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Iclaprim — Experimental treatment
  Other Names: MTF-100
  Arms: iclaprim
Drug: Vancomycin — Active comparator
  Other Names: Vancocin
  Arms: vancomycin

SUMMARY:
This is a multicenter, randomized, double-blind study of the efficacy and safety of iclaprim compared to vancomycin for the treatment of skin and skin structure infections.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind study of the efficacy and safety of IV iclaprim compared to IV vancomycin. Patients will receive either iclaprim or vancomycin for 5 to 14 days. Patients will be evaluated daily up to early time point (ETP), then every 48 to 72 hours through the end of treatment. Patients will also be evaluated at the test of cure (TOC) visit (7 to 14 days post-EOT), and will have a Late Follow-Up (LFU) visit (28 to 32 days post-first dose).

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent;
2. ≥18 years of age;
3. a bacterial infection of the skin with a lesion size area of at least 75 cm2;
4. a major cutaneous abscess, cellulitis/erysipelas, and/or wound infections;
5. the presence of purulent or seropurulent drainage or at least three signs and symptoms of infection (discharge, erythema, swelling, warmth, or pain).

Exclusion Criteria:

1. severely impaired arterial blood supply such that amputation of the infected anatomical site is likely;
2. infected diabetic foot ulcers;
3. infected decubitus ulcers;
4. necrotizing fasciitis or gangrene;
5. uncomplicated skin or skin structure infection;
6. infections associated with a prosthetic device;
7. suspected or confirmed osteomyelitis;
8. conditions requiring systemic anti-microbial treatment, prophylaxis, or suppression therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2015-11; Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Noviello, MD, Study Director — Motif Biosciences
Locations (47):
- United States (16):
  - California, Anaheim, California
  - California, Buena Park, California
  - California, Chula Vista, California
  - California, La Palma, California
  - California, Long Beach, California
  - St. Mary Medical Center ER, Long Beach, California
  - Florida, Hollywood, Florida
  - Florida, Miami, Florida
  - Georgia, Columbus, Georgia
  - Montana, Butte, Montana
  - Nevada, Las Vegas, Nevada
  - New Jersey, Somers Point, New Jersey
  - Ohio, Lima, Ohio
  - Tennessee, Smyrna, Tennessee
  - Washington, Kennewick, Washington
  - Washington, Richland, Washington
- Argentina, Buenos Aires, Argentina
- Belgium, Brussels, Belgium
- Croatia (3):
  - Croatia, Slavonski Brod
  - Croatia, Zadar
  - Croatia, Zagreb
- Czechia (4):
  - Czech Republic, Hradec Králové
  - Czech Republic, Ostrava
  - Czech Republic, Příbram
  - Czech Republic, Ústí nad Labem
- Estonia (4):
  - Estonia, Kohtla-Järve
  - Estonia, Tallinn
  - Estonia, Tartu
  - Estonia, Võru
- Hungary (5):
  - Hungary, Budapest
  - Hungary, Miskolc
  - Hungary, Szeged
  - Hungary, Székesfehérvár
  - Hungary, Veszprém
- Portugal (5):
  - Portugal, Amadora
  - Portugal, Braga
  - Portugal, Porto
  - Portugal, Santarém
  - Portugal, Viana do Castelo
- Romania (5):
  - Romania, Arad
  - Romania, Bucharest
  - Romania, Cluj-Napoca
  - Romania, Craiova
  - Romania, Timișoara
- Turkey (Türkiye) (3):
  - Turkey, Aydin
  - Turkey, Istanbul
  - Turkey, Trabzon

REFERENCES:
- [Derived] Huang DB, Corey GR, Holland TL, Lodise T, O'Riordan W, Wilcox MH, File TM Jr, Dryden M, Balser B, Desplats E, Torres A. Pooled analysis of the phase 3 REVIVE trials: randomised, double-blind studies to evaluate the safety and efficacy of iclaprim versus vancomycin for treatment of acute bacterial skin and skin-structure infections. Int J Antimicrob Agents. 2018 Aug;52(2):233-240. doi: 10.1016/j.ijantimicag.2018.05.012. Epub 2018 May 19. PMID 29783024
- [Derived] Holland TL, O'Riordan W, McManus A, Shin E, Borghei A, File TM Jr, Wilcox MH, Torres A, Dryden M, Lodise T, Oguri T, Corey GR, McLeroth P, Shukla R, Huang DB. A Phase 3, Randomized, Double-Blind, Multicenter Study To Evaluate the Safety and Efficacy of Intravenous Iclaprim versus Vancomycin for Treatment of Acute Bacterial Skin and Skin Structure Infections Suspected or Confirmed To Be Due to Gram-Positive Pathogens (REVIVE-2 Study). Antimicrob Agents Chemother. 2018 Apr 26;62(5):e02580-17. doi: 10.1128/AAC.02580-17. Print 2018 May. PMID 29530858

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Iclaprim | Vancomycin
Started | 306 | 307
Completed | 295 | 305
Not Completed | 11 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iclaprim | Vancomycin | Total
Number analyzed (Participants) | 295 | 305 | 600
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 240 | 250 | 490
  >=65 years | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (15.7) | 50.8 (15.0) | 50.4 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 108 | 211
  Male | 192 | 197 | 389
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 99 | 94 | 193
  Not Hispanic or Latino | 193 | 207 | 400
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 12 | 11 | 23
  White | 267 | 276 | 543
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 12 | 9 | 21
Region of Enrollment [Number; unit: participants]
  Argentina | 9 | 3 | 12
  Romania | 20 | 14 | 34
  Turkey | 5 | 7 | 12
  Belgium | 2 | 0 | 2
  Hungary | 4 | 5 | 9
  United States | 200 | 205 | 405
  Czechia | 4 | 3 | 7
  Portugal | 3 | 5 | 8
  Estonia | 36 | 48 | 84
  Croatia | 10 | 12 | 22
  Mexico | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With ≥20% Reduction in Lesion Size at 48 to 72 Hours Compared to Baseline
Description: ≥20% reduction in lesion size at 48 to 72 hours (Early Time Point [ETP]) compared to baseline in all randomized patients (ITT).
Time Frame: Baseline and 48 to 72 hours after first dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Iclaprim | Vancomycin
Number analyzed (Participants) | 295 | 305
percentage of participants | 78.3 [73.2 to 82.9] | 76.7 [71.6 to 81.3]

2. Secondary Outcome: Number of Participants With Resolution or Near Resolution of Lesion at Test of Cure Visit
Description: Resolution or Near Resolution of Lesion at Test of Cure (TOC) Visit.
Time Frame: 7 to14 days after the end of treatment
Measure: Number; unit: participants
Arm/Group | Iclaprim | Vancomycin
Number analyzed (Participants) | 295 | 305
participants | 229 | 237

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Iclaprim | Vancomycin
All-Cause Mortality (participants affected / at risk) | 0/299 | 1/302
Serious Adverse Events (participants affected / at risk) | 0/299 | 1/302
Other Adverse Events (participants affected / at risk) | 0/299 | 1/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iclaprim (N=299) | Vancomycin (N=302)
Renal and urinary disorders (Renal and urinary disorders) | 0 | 1 — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iclaprim (N=299) | Vancomycin (N=302)
Product Issues (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2015-12-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT02607618/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT02607618/SAP_001.pdf